CLINICAL TRIAL: NCT07024160
Title: A Single-center, Randomized, Double-blind, Placebo-controlled Phase I Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Dose (SAD) Administration of MT1011 Injection in Healthy Subjects
Brief Title: Phase I Study of MT1011 Injection in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT1011-I-C02
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-05

CONDITIONS: Used in Patients Receiving Anticoagulant Therapy (e.g., Rivaroxaban or Apixaban, Inhibitors of Coagulation Factor Xa) Who Require Reversal of Anticoagulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MT1011 (Experimental): Interventional: The SAD study involves single administration of MT1011
  Interventions: Drug: MT1011
- Placebo (Placebo Comparator): Placebo: The SAD study involves single administration of Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT1011 — MT1011 is a novel synthetic small molecule anticoagulant reversal agent for reversing anticoagulant effects including factor IIa and Xa inhibitors.
  Arms: MT1011
Drug: Placebo — This intervention contains no active ingredients
  Arms: Placebo

SUMMARY:
This is a single-center, randomized,double-blind, placebo-controlled Phase I study to evaluate safety, PK and PD of single ascending dose (SAD) of MT1011 injection in healthy adult subjects. Includes 5 dose cohorts, with 40 subjects planned for enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects (with at least 1/4 being either female or male), aged 18 to 45 years (inclusive) at screening;
2. Body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females at screening, with a Body Mass Index [BMI = weight (kg) / height² (m²)] within the range of 18.5 to 26.0 kg/m² (inclusive);
3. Subjects must provide informed consent for this study prior to participation and voluntarily sign a written informed consent form;
4. Subjects must be able to maintain good communication with the investigators.

Exclusion Criteria:

1. Subjects with abnormal and clinically significant findings in vital signs, physical examination, laboratory tests (blood routine, urinalysis, blood biochemistry, coagulation function), abdominal ultrasound, or chest X-ray as determined by the investigator;
2. Women who are pregnant or breastfeeding, or female subjects with positive pregnancy tests; Subjects (or their partners) planning pregnancy, or planning to donate sperm/ova during the study or within

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of AEs (Adverse Events) and SAEs (Serious Adverse Events)and treatment-related adverse events (TEAEs). | up to Day 14
  The occurrence of all adverse events (AEs), serious adverse events (SAEs)

SECONDARY OUTCOMES:
Cmax of MT1011 | Within 1 hour before dosing on Day 1 (D1), and at 5min,15min,0.5,1, 2, 4, 8, 12, 24, 48 hours post-dose.
  Cmax - Maximum plasma concentration
Tmax of MT1011 | Within 1 hour before dosing on Day 1 (D1), and at 5min,15min,0.5,1, 2, 4, 8, 12, 24, 48 hours post-dose.
  Tmax - Time to reach Cmax
T1/2 of MT1011 | Within 1 hour before dosing on Day 1 (D1), and at 5min,15min,0.5,1, 2, 4, 8, 12, 24, 48 hours post-dose.
  t1/2 - Elimination half-life
AUC0-tau of MT1011 | Within 1 hour before dosing on Day 1 (D1), and at 5min,15min,0.5,1, 2, 4, 8, 12, 24, 48 hours post-dose.
  AUC0-tau - Area under the plasma concentration-time curve during one dosing interval
AUC0-t of MT1011 | Within 1 hour before dosing on Day 1 (D1), and at 5min,15min,0.5,1, 2, 4, 8, 12, 24, 48 hours post-dose.
  AUC0-t - Area under the plasma concentration-time curve from time zero to the last measurable concentration
Whole blood clotting time | Within 1 hour before dosing on Day 1 (D1), and at 15min, 2, 24 hours post-dose.
  Whole blood clotting time
Activated partial thromboplastin time | Within 1 hour before dosing on Day 1 (D1), and at 15min, 2, 24 hours post-dose.
  Activated partial thromboplastin time
Prothrombin time | Within 1 hour before dosing on Day 1 (D1), and at 15min, 2, 24 hours post-dose.
  Prothrombin time
fibrinogen | Within 1 hour before dosing on Day 1 (D1), and at 15min, 2, 24 hours post-dose.
  fibrinogen
International normalized ratios | Within 1 hour before dosing on Day 1 (D1), and at 15min, 2, 24 hours post-dose.
  International normalized ratios
Thrombin time | Within 1 hour before dosing on Day 1 (D1), and at 15min, 2, 24 hours post-dose.
  Thrombin time
Factor Xa activity | Within 1 hour before dosing on Day 1 (D1), and at 15min, 2, 24 hours post-dose.
  Factor Xa activity

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality, China